CLINICAL TRIAL: NCT05589896
Title: A First-in-Human Study of HLA-Partially to Fully Matched Allogenic Cryopreserved Deceased Donor Bone Marrow Transplantation for Patients With Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ossium Health, Inc. (Industry)
Collaborators: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRESERVE I
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Acute Biphenotypic Leukemia; Acute Undifferentiated Leukemia; CLL (Chronic Lymphocytic Leukemia); Chronic Myeloid Leukemia (CML); MDS (Myelodysplastic Syndrome); Non-Hodgkin Lymphomas; Hodgkins Lymphoma; Cutaneous T Cell Lymphomas (CTCL)
Keywords: Leukemia; Hematologic Diseases; ALL; AML; ABL; AUL; Bone Marrow Transplant; Lymphoma; MDS; CLL; CML
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Leukemia; Hematologic Diseases; Lymphoma | interventions — Bone Marrow Transplantation; fludarabine phosphate; Cyclophosphamide; Mesna; Melphalan; Mycophenolic Acid; Filgrastim

STUDY DESIGN:
Intervention Model Description: All patients will receive Ossium HPC, Marrow product. Study arms will be based on order of enrollment and planned conditioning regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Bone Marrow Transplant with Ossium HPC, Marrow
  Pre-transplant myeloablative conditioning treatment with:
  Regimen A(MAC): Busulfan and Fludarabine
  [OR]
  Regimen B(MAC): Fludarabine and Total Body Irradiation
  [OR]
  Regimen C(RIC): Fludarabine, Cyclophosphamide, and Total Body Irradiation
  [OR]
  Regimen D (RIC): Fludarabine, Melphalan, and Total Body Irradiation
  Post-Transplant treatment with Cyclophosphamide, Tacrolimus, Mycophenolate Mofetil, and Filgrastim
  Interventions: Other: Ossium HPC Marrow, Bone Marrow Transplant; Other: Pre-transplant conditioning - Myeloablative (MAC); Other: Pre-transplant conditioning - Reduced Intensity (RIC); Other: Post-transplant treatment
- Cohort 2 (Experimental): *Open to enrollment after DSMB review of Cohort 1 safety events through Day 56*
  Bone Marrow Transplant with Ossium HPC, Marrow
  Pre-transplant conditioning treatment with:
  Regimen A(MAC): Busulfan and Fludarabine
  [OR]
  Regimen B(MAC): Fludarabine and Total Body Irradiation
  [OR]
  Regimen C(RIC): Fludarabine, Cyclophosphamide, and Total Body Irradiation
  [OR]
  Regimen D(RIC): Fludarabine, Melphalan, and Total Body Irradiation
  Post-Transplant treatment with Cyclophosphamide, Tacrolimus, Mycophenolate Mofetil, and Filgrastim
  Interventions: Other: Ossium HPC Marrow, Bone Marrow Transplant; Other: Pre-transplant conditioning - Myeloablative (MAC); Other: Pre-transplant conditioning - Reduced Intensity (RIC); Other: Post-transplant treatment

INTERVENTIONS:
Other: Ossium HPC Marrow, Bone Marrow Transplant — Hematopoetic Cell Transplantation
Other: Pre-transplant conditioning - Myeloablative (MAC) — Regimen A or Regimen B
  Other Names: Busuflex; Fludara; TBI
Other: Pre-transplant conditioning - Reduced Intensity (RIC) — Regimen C or Regimen D
  Other Names: Fludara; Cytoxan; Mesnex; TBI; Melphalan
Other: Post-transplant treatment — Post-transplant treatment
  Other Names: Cytoxan; Mesnex; CellCept; Filgrastim

SUMMARY:
The goal of this clinical trial is to determine the safety and feasibility of allogeneic transplantation with bone marrow from a deceased donor in patients with acute and chronic leukemias, myelodysplastic syndrome, and certain lymphomas. Patients will either receive myeloablative conditioning or reduced intensity conditioning regimen prior to the transplant. Patients will be followed for 56 days for safety endpoints and remain in follow-up for one year.

ELIGIBILITY:
Inclusion Criteria:

* Patient has the ability to provide informed consent according to the applicable regulatory and local institutional requirements
* Male or female, aged ≥18 and ≤65 years for patients receiving MAC (Regimen A or Regimen B); aged ≥18 and ≤75 years for patients receiving RIC (Regimen C or D)
* Patient must require allogeneic HCT per the discretion of the treating physician
* Patient must be high-resolution, HLA partially or fully matched (4-8/8 allele matched at HLA-A, -B, -C, DRB1) to an available Ossium HPC, Marrow product
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosed with malignant hematologic disease including:

  1. Acute leukemia [acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML), acute biophenotypic leukemia (ABL), or acute undifferentiated leukemia (AUL)], MDS without fibrosis, or chronic leukemia (CLL, CML) in the first remission or beyond with ≤5% marrow blasts documented by bone marrow assessment and no circulating blasts or extra-medullary disease within 42 days prior to anticipated start of conditioning
  2. Chemosensitive non-Hodgkin's lymphomas, Hodgkin's lymphoma, or cutaneous T cell lymphomas in the first remission or beyond documented by PET/CT imaging and bone marrow assessment within 42 days prior to anticipated start of conditioning
* Karnofsky performance status score ≥70% (MAC) or ≥60% (RIC)
* HCT comorbidity index (HCT-CI) ≤5
* Adequate organ function defined as:

  1. Cardiac: LVEF at rest ≥40% (RIC) or LVEF at rest ≥45% (MAC)
  2. Pulmonary: DLCO, FEV1, FVC ≥50% predicted by pulmonary function tests (PFTs). DLCO value may be corrected for hemoglobin.
  3. Hepatic: total bilirubin ≤2.0 mg/dL, and ALT, AST, and ALP <3 x upper limit normal (ULN), unless ALT, AST, and/or ALP are disease related
  4. Renal: SCr within 1.5x normal range for age. If SCr is outside normal range for age, CrCl> 60 mL/min/1.73m2 must be obtained (measured by 24-hour urine specimen or nuclear glomerular filtration rate (GFR), or calculated GFR)

Exclusion Criteria:

* Availability of suitable graft from living donor (defined as 7/8 or 8/8 HLA-matched related or unrelated donors, haploidentical donors, or cord blood donors)
* Prior autologous or allogeneic HCT
* Pregnancy or lactation
* Ongoing treatment with an investigational drug used for disease-related treatment within 5 half-lives of the drug
* Current uncontrolled bacterial, viral or fungal infection defined as currently taking medication with evidence of progression of clinical symptoms or radiologic findings
* Any condition(s) or diagnosis, both physical or psychological, or physical exam finding that in the investigator's opinion precludes participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Engraftment | Day 28
  Neutrophil engraftment is defined as achieving an absolute neutrophil count (ANC) of greater than or equal to 500/µL for 3 consecutive measurements on 3 different days by Day 28.
Serious Adverse Events | Day 56
  Occurrence of any event classified as SAE. The time of occurrence of each serious adverse event will be recorded.
CTCAE Grade 3/4 Adverse Events (AEs) | Day 56
  Occurrence of any event classified as grade 3/4 AE attributed to Ossium HPC, Marrow per the CTCAE v5.0 guidelines. The time of the occurrence of each event will be recorded.
CTCAE Grade 3/4 Adverse Events (AEs) attributed to infusion of Ossium HPC, Marrow | Day 28
  Occurrence of any event classified as grade 3 or higher attributed to Ossium HPC, Marrow infusion per the CTCAE v5.0 guidelines. The time of the occurrence will be recorded.
Death | Day 56
  The time of death will be recorded for each expired patient.

SECONDARY OUTCOMES:
Cumulative incidences of neutrophil engraftment | Day 28
  Neutrophil engraftment in defined as achieving an absolute neutrophil count (ANC) of greater than or equal to 500/µL for 3 consecutive measurements on different days by Day 28.
Cumulative incidences of platelet recovery | Day 56
  Platelet recovery is defined as platelets greater than or equal to 20,000/µL for 3 consecutive days in the absence of transfusion for 7 consecutive days by Day 56.
Cumulative incidence of disease relapses | Day 365
  The cumulative incidence of relapse is measured from the date of transplant (Day 0) until the date of relapse or progression; patients not known to have relapsed are censored on the date they were last examined; patients who died without relapse are counted as a competing cause of failure.
Transplant-related mortality (TRM) | Day 100 and Day 365
  TRM is defined as death without evidence of disease progression or recurrence.
Cumulative incidences of acute (aGVHD) Graft Versus Host Disease | Day 100, Day 180, and Day 365
  aGVHD is defined as any skin, gastrointestinal or liver abnormalities fulfilling the criteria of grades II-IV or grades III-IV.
Cumulative incidences of chronic (cGVHD) Graft Versus Host Disease | Day 100, Day 180, and Day 365
  cGVHD is defined per National Institutes of Health (NIH) Consensus Criteria and includes organ involvement and severity, and overall global composite score (mild/moderate/severe).
Incidence of clinically-significant infections | Day 100 and Day 365
  A clinically significant infection is defined as any microbiologic or radiographic infection for which antimicrobial therapy was administered.

OTHER OUTCOMES:
Length of Stay in Hospital | Day 100 and Day 365
  Cumulative days alive and out of the hospital in the first 100 days and in the first year post-transplant.
Time to provide Ossium product to the patient from product availability request | Day 365
  Time from preliminary search to find a donor match in the Ossium registry and the time to provide Ossium HPC, Marrow product to recipient (time from donor availability request to delivery of product to transplant center).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Auletta, MD, Study Chair — Center for International Blood and Marrow Transplant Research
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Columbia University - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - TriStar Bone Marrow Transplant, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Methodist Hospital, Texas Transplant, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No